CLINICAL TRIAL: NCT00005838
Title: Multicenter, Open-Ended, Double-Blind, Placebo-Controlled, Phase III Study of AE-941 in Addition to Combined Modality Treatment (Chemotherapy/Radiotherapy) for Locally Advanced Unresectable Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy Plus Radiation Therapy With or Without AE-941 in Treating Patients With Stage III Non-small Cell Lung Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02725; ID99-303; U10CA045809 (NIH); CDR0000067853 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Lung; Adenosquamous Cell Lung Cancer; Large Cell Lung Cancer; Squamous Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — shark cartilage extract; Cisplatin; Vinorelbine; Carboplatin; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (shark cartilage extract AE-941) (Experimental): Patients receive oral AE-941 (Neovastat) twice daily beginning on day 1 or within 10 days of initiation of chemotherapy.
  All patients receive induction chemotherapy with 1 of the following platinum-based regimens: cisplatin IV on days 1, 22, 50, and 71 and vinorelbine IV on days 1, 8, 22, 29, 50, 57, 71, and 78 carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on days 1, 22, 50, 57, 64, 71, 78, and 85.
  All patients receive radiotherapy beginning on day 50 for 6 weeks. Treatment in both arms continues in the absence of unacceptable toxicity.
  Interventions: Drug: shark cartilage extract AE-941; Drug: cisplatin; Drug: vinorelbine tartrate; Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo twice daily beginning on day 1 or within 10 days of initiation of chemotherapy.
  All patients receive induction chemotherapy with 1 of the following platinum-based regimens: cisplatin IV on days 1, 22, 50, and 71 and vinorelbine IV on days 1, 8, 22, 29, 50, 57, 71, and 78 carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on days 1, 22, 50, 57, 64, 71, 78, and 85.
  All patients receive radiotherapy beginning on day 50 for 6 weeks. Treatment in both arms continues in the absence of unacceptable toxicity.
  Interventions: Other: placebo; Drug: cisplatin; Drug: vinorelbine tartrate; Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: shark cartilage extract AE-941 — Given orally
  Other Names: AE-941; Neovastat; Neovastat/AE-941
  Arms: Arm I (shark cartilage extract AE-941)
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells. AE-941 may help shrink or slow the growth of non-small cell lung cancer cells. It is not yet known if combination chemotherapy plus radiation therapy is more effective with or without AE-941 for non-small cell lung cancer. This randomized phase III trial is studying combination chemotherapy and radiation therapy given with AE-941 to see how well they work compared to combination chemotherapy and radiation therapy alone in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall survival of patients with unresectable stage IIIA or IIIB non-small cell lung cancer treated with induction platinum-based chemotherapy and radiotherapy with or without AE-941 (Neovastat).

II. Determine the progression-free survival, tumor response, tumor response duration, and metastasis-free survival of patients treated with these regimens.

III. Determine the tolerability of this regimen in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to stage (IIIA vs IIIB), type of platinum-based induction chemotherapy to be received (cisplatin and vinorelbine vs carboplatin and paclitaxel), and gender. Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive oral AE-941 (Neovastat) twice daily beginning on day 1 or within 10 days of initiation of chemotherapy.

Arm II: Patients receive oral placebo twice daily beginning on day 1 or within 10 days of initiation of chemotherapy.

All patients receive induction chemotherapy with 1 of the following platinum-based regimens: cisplatin IV on days 1, 22, 50, and 71 and vinorelbine IV on days 1, 8, 22, 29, 50, 57, 71, and 78 carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on days 1, 22, 50, 57, 64, 71, 78, and 85.

All patients receive radiotherapy beginning on day 50 for 6 weeks. Treatment in both arms continues in the absence of unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 756 patients (378 per treatment arm) will be accrued for this study within 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed newly diagnosed, untreated, unresectable stage IIIA or stage IIIB non-small cell lung cancer

  * Squamous cell carcinoma, adenocarcinoma, or large cell carcinoma of the lung
  * Mixed tumors allowed if non-small cell elements identified
  * Contralateral supraclavicular and/or scalene lymph node involvement allowed
  * No disease extending into the cervical region
* At least 1 bidimensionally or unidimensionally measurable lesion
* No pleural effusion unless cytologically negative or too small to safely aspirate
* Not scheduled for curative cancer surgery
* Performance status - ECOG 0-1
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hematocrit greater than 30%
* SGOT or SGPT less than 1.5 times upper limit of normal
* Bilirubin normal
* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min
* No other major medical or psychiatric illness that would preclude study participation or consent
* No medical condition that interferes with oral medication intake and/or absorption (gastrectomy or major intestinal resection)
* No grade 2 or greater peripheral neuropathy unless secondary to mechanical etiology
* No hypersensitivity to fish products
* No more than 10% weight loss within past 3 months
* No other malignancy within past 3 years except inactive carcinoma in situ of the cervix or nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 30 days since prior chemotherapy
* See Disease Characteristics
* Recovered from prior major surgery
* At least 30 days since prior shark cartilage products
* No other concurrent investigational anticancer agents
* No other concurrent cartilage products
* No other concurrent investigational agents
* No concurrent amifostine or other radioprotectants
* No concurrent enrollment in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2000-03; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | From randomization until date of death or last follow-up, assessed up to 7 years
  Survival distributions will be compared by use of the log-rank test. The stratified log-rank test (nominal or categorical covariates) may be used to simultaneously control for important prognostic factors. Kaplan-Meier curves will also be plotted to illustrate the comparative survival experience of both groups over the entire study period.

SECONDARY OUTCOMES:
Progression-free survival every 3 months | From randomization until disease progression, assessed up to 7 years
  Will be compared by use of the log-rank test. The stratified log-rank test (nominal or categorical covariates) may be used to simultaneously control for important prognostic factors. Kaplan-Meier curves will also be plotted.
Tumor response rate | Up to 7 years
  Will be compared by chi-square test.
Tumor response duration | From first observation of at least a partial response to detection of disease progression or death due to any cause, assessed up to 7 years
  Will be compared by use of the log-rank test. The stratified log-rank test (nominal or categorical covariates) may be used to simultaneously control for important prognostic factors. Kaplan-Meier curves will also be plotted.
Metastasis-free survival | From randomization until metastasis documented by imaging procedures, assessed up to 7 years
  Will be compared by use of the log-rank test. The stratified log-rank test (nominal or categorical covariates) may be used to simultaneously control for important prognostic factors. Kaplan-Meier curves will also be plotted.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States